CLINICAL TRIAL: NCT00591214
Title: A Phase I, Open-Label, Single-Dose Study of MP-424 in Patients With Genotype 1b Hepatitis C
Brief Title: Safety and PK Study of MP-424 to Treat Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: G060-A3
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Protease Inhibitor
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP-424 (Experimental)
  Interventions: Drug: MP-424 (Telaprevir)

INTERVENTIONS:
Drug: MP-424 (Telaprevir) — Three tablets of MP-424 250mg tablet at a time, every 8 hours, 12 weeks administration (dose in a day: 2250 mg)

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and HCV(Hepatitis C virus) RNA (Ribonucleic Acid) kinetics after administration of MP-424 to patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with genotype 1b chronic hepatitis C
* Patients naive to the concomitant medications with interferon

Exclusion Criteria:

* Patients diagnosed with decompensated cirrhosis
* Patients diagnosed with positive HBs(Hepatitis B virus surface) antigen in the test

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fumitaka Suzuki, MD, Principal Investigator — Department of Hepatology, Toranomon Hospital
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Yamada I, Suzuki F, Kamiya N, Aoki K, Sakurai Y, Kano M, Matsui H, Kumada H. Safety, pharmacokinetics and resistant variants of telaprevir alone for 12 weeks in hepatitis C virus genotype 1b infection. J Viral Hepat. 2012 Feb;19(2):e112-9. doi: 10.1111/j.1365-2893.2011.01514.x. Epub 2011 Oct 7. PMID 22239508

RESULTS

PARTICIPANT FLOW:
Groups:
- MP-424: Drug: MP-424 750 mg every 8 hours for 12 weeks Other Name: Telaprevir
Period: Overall Study
Arm/Group | MP-424
Started | 10
Completed | 2
Not Completed | 8
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MP-424
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration in Plasma) of MP-424
Description: Date were collected at Day1 (0 (pre-dose), 1 ,2.5, 4, 6, 8, 12, 16 hours post-dose), Day14 (0 (pre-dose), 1, 2.5, 4, 6, 8, 12, 16 hours post-dose) and Day85 (0 (pre-dose), 1, 2.5, 4, 6, 8, 12, 16, 24 hours post-dose). Date as pre-dose were collected at Day2, Day3, Day8, Day15, Day29, Day43 and Day57.
Time Frame: Date were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: μg / mL
Arm/Group | MP-424
Number analyzed (Participants) | 10
μg / mL
  Day 1 (10 cases) | 2.24 (0.93)
  Day 14 (10 cases) | 3.34 (1.11)
  Day 85 (3 cases) | 3.68 (1.29)

2. Primary Outcome: Tmax (Time of Maximum Plasma Concentration) of MP-424
Description: as for outcome 1
Time Frame: Date were collected at Day1 to Day85
Measure: Median (Full Range); unit: hours
Arm/Group | MP-424
Number analyzed (Participants) | 10
hours
  Day 1 (10 cases) | 2.50 [2.30 to 7.92]
  Day 14 (10 cases) | 2.49 [0.98 to 5.97]
  Day 85 (3 cases) | 2.72 [2.68 to 4.00]

3. Primary Outcome: AUC 0-8h (Area Under the Concentration-time Curve From Time Zero to 8 Hours) of MP-424
Description: as for outcome 1
Time Frame: Date were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: μg x h /mL
Arm/Group | MP-424
Number analyzed (Participants) | 10
μg x h /mL
  Day 1 (10 cases) | 11.60 (4.74)
  Day 14 (10 cases) | 22.31 (8.29)
  Day 85 (3 cases) | 23.98 (9.45)

4. Primary Outcome: Ctrough (Plasma Trough Concentration) of MP-424
Description: as for outcome 1
Time Frame: Date were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MP-424
Number analyzed (Participants) | 10
μg/mL
  Day1 (10 cases) | 1.462 (0.949)
  Day 14 (10 cases) | 2.239 (0.953)
  Day 85 (3 cases) | 2.312 (1.265)

5. Primary Outcome: t1/2 (Half Life Period) of MP-424
Description: as for outcome 1
Time Frame: Date were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MP-424
Number analyzed (Participants) | 10
hours
  Day 1 (7 cases) | 5.57 (2.67)
  Day 14 (8 cases) | 9.64 (6.14)
  Day 85 (3 cases) | 18.35 (22.91)

6. Secondary Outcome: Change in HCV RNA Levels of MP-424
Description: Date were collected at Day -28, Day1 (0 (pre-dose), 2.5, 4, 8, 16 hours post-dose), Day2, Day3, Day8, Day14, Day29, Day43, Day57, Day86.
  Change Value was calculated as the each time point minus the baseline point which was averaged Day -28 and Day0-0hour(pre-dose)).
Time Frame: Day1 (2.5, 4, 8, 16 hours), Day2, Day3, Day8, Day14, Day29, Day43, Day57 and Day86
Measure: Mean (Standard Deviation); unit: Log IU / mL
Arm/Group | MP-424
Number analyzed (Participants) | 10
Log IU / mL
  Day 1_2.5h (9 cases) | 0.100 (0.217)
  Day 1_4h (10 cases) | -0.195 (0.207)
  Day 1_8h (10 cases) | -1.115 (0.376)
  Day 1_16h (10 cases) | -2.435 (0.408)
  Day 2 before dosing (10 cases) | -2.955 (0.323)
  Day 3 (10 cases) | -3.735 (0.369)
  Day 8 (10 cases) | -4.505 (0.633)
  Day 14 (10 cases) | -4.895 (0.675)
  Day 29 (10 cases) | -4.785 (1.203)
  Day 43 (10 cases) | -3.815 (1.344)
  Day 57 (5 cases) | -4.120 (2.086)
  Day 86 (3 cases) | -3.867 (2.363)

ADVERSE EVENTS:
Arm/Group | MP-424
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=10)
Nasopharyngitis (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 2
Malaise (General disorders) | 2
Thirst (General disorders) | 1
Low density lipoprotein increased (Investigations) | 5
Blood uric acid increased (Investigations) | 5
Blood triglycerides increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood luteinising hormone increased (Investigations) | 1
Eosinophil percentage increased (Investigations) | 1
Lymphocyte percentage decreased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Palpitation (Cardiac disorders) | 1
Conjunctivitis (Eye disorders) | 1
Myodesopsia (Eye disorders) | 1
Ginginal swelling (Gastrointestinal disorders) | 1
Blood gonadotropin increased (Investigations) | 1
Differential white blood cell count abnormal (Investigations) | 1
Facial palsy (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other